CLINICAL TRIAL: NCT02921178
Title: Effects of Omalizumab Compared to Non-Omalizumab Treatment in the Propensity- Matched Group on Asthma Exacerbation in Asthma Patients in Korea: a Retrospective Cohort in a Real World
Brief Title: Effects of Omalizumab Compared to Non-Omalizumab Treatment in Asthma Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Hae-Sim Park, Ajou University Hospital, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-MDB-16-276
Record Dates: First submitted 2016-09-22; First posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Omalizumab — comparision of using Omalizumab and non-Omalizumab treatment
  Other Names: Xolair

SUMMARY:
The purpose of this study is effects of Omalizumab compared to non-Omalizumab treatment in the propensity-matched group on asthma exacerbation in asthma patients in Korea: a retrospective cohort in real world.

Omalizumab was approved 2007 in Korea and has been used in this center. We would like to collect and analyze the data and exacerbation outcomes of these patients on Omalizumab; no Korean real world data available.

DETAILED DESCRIPTION:
1. Primary and secondary outcomes and analysis methods

(1) Primary endpoint Comparison of asthma exacerbation rates of omalizumab-treated vs non-Omalizumab treated group at outcome period (6 months). (asthma exacerbation: at least 1 systemic steroid treatment and/or bursts of systemic oral steroid use by prednisone-equivalent dose ≥45mg/3days, in a 6 month for relieving asthma exacerbations.) Fisher's exact test is examined for asthma exacerbation between omalizumab-treated vs non-Omalizumab treated group.

(2) Secondary endpoint

* Comparison of the clinical parameters Asthma exacerbation rate, ICS sparing effect, OCS requirement, lung function (FEV1%), Healthcare resource use (asthma-related ER visit/hospitalization)

  1. Within Omalizumab-treated group between baseline and outcome period
  2. Between Omalizumab-treated and not-treated groups at outcome period For comparison of within group, paired T-test and McNemar test are applied for continuous and categorical parameters, respectively. And, T-test and Fisher's exact test are examined for continuous and categorical parameters between Omalizumab-treated and not-treated groups. Incidentally, non-parametric tests will be examined as needed.
* Finding predictor of favorable responders to Omalizumab at 6 months. (Favorable responder: 50% reduction of asthma exacerbation or of steroid requirement during 6 months with/without ICS/LABA) Candidate factors: Omalizumab treatment period/monthly dose, age, gender, asthma treatment duration, total IgE, sputum cell profile, peripheral eosinophilia serum periostin level, anti-asthmatic drug requirements etc.

Binary logistic regression is used for finding predictor of favorable responders. If a serious imbalance of dependent parameter occurs from a low frequency of favorable responder, the descriptive analysis will be applied with T-test and Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

1. Codes for asthma (ICD-10: J45) dependent on availability

   * Who have been diagnosed as having allergic asthma with asthma exacerbations (J45 asthma, J45.0 predominantly allergic asthma and J45.8 mixed asthma)
   * Those who initially diagnosed as J45.9 asthma, unspecified, we will refer the evidence of allergic components such as IgE level and skin prick test result.
2. Aged 18-80 years at index date
3. Active asthma, defined as ≥ 1 prescriptions for LABA/ICS during baseline periods
4. un-controlled asthma during the baseline period Any one of three criteria A. Asthma exacerbation B. Asthma-related ER visit/Hospitalization C. Physician defined un-controlled asthma

   * Worsening symptom status
   * Worsens on tapering of high dose ICS or systemic CS
   * Air flow limitation (after appropriate bronchodilator withhold FEV1%<80% predicted)

Exclusion Criteria:

* taken biologics during baseline and outcome period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult asthmatic patients(Duration of accumulated data electronic medical records)
Sampling Method: Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
asthma exacerbation rate | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hae-sim Park, Ph.D., Principal Investigator — Ajou University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided